CLINICAL TRIAL: NCT01854502
Title: Organizing Family-based Health Promotion for Young Children in Public Dental Service
Brief Title: Family-based Counseling Models for Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Irma Arpalahti, chief dentist, University of Turku
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IArpalahti2008
Record Dates: First submitted 2013-05-03; First posted 2013-05-15 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Dental Plaque; Dental Caries; Behaviorial Habits
Keywords: Young children; counseling; fluoride; xylitol
MeSH Terms: conditions — Dental Plaque; Dental Caries; Habits | interventions — Oral Hygiene; Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oral hygiene and fluoride use (Experimental): Parents of young children were given counseling of their own oral hygiene and the use of fluoride on their child's visit to public dental service. The child was given multi-faceted counseling for good oral health habits.
  Interventions: Behavioral: Oral hygiene and fluoride use
- Control (No Intervention): Control, The parents were not given any intervention on their child's visit to public dental service.
  The child was given multi-faceted counseling for good oral health habits.
- Diet and use of xylitol (Experimental): Parents of young children were given counseling of their own diet and the use of xylitol on their child's visit to public dental service. The child was given multi-faceted counseling for good oral health habits.
  Interventions: Behavioral: Diet and use of xylitol

INTERVENTIONS:
Behavioral: Oral hygiene and fluoride use — Parents were given instructions how to brush and clean between teeth and to use fluoride toothpaste two times a day.
  Arms: Oral hygiene and fluoride use
Behavioral: Diet and use of xylitol — Parents were asked to fill in one-day diaries of their own diet in the waiting room. The dental professional pointed out the frequency of meals and snacks, as well as suggested the timing of xylitol products.
  Arms: Diet and use of xylitol

SUMMARY:
The purpose of this study is to compare the effects of two new family-based oral health promotion programs with the routine program in use earlier in Vantaa public dental service. The children born in 2008 were followed from their first visit to public dental service at the age of 6-12 months to their dental examination at the age of 2-2½ years. The outcome measures are the colonization of mutans streptococci in dental plaque, dental caries, and the oral health habits of two-year-olds.

DETAILED DESCRIPTION:
The investigators hypothesized that the training of the dental professionals involved in children's examinations could improve the quality of the counseling, raise the level of commitment, and give them a new kind of perspective on early childhood oral health counseling. Health promotion programs with clinical guidance aimed also at the parents themselves might commit the families to maintain their children's good oral health.

All programs (two new and the control program) consisted of the basic elements of oral health counseling for the children. The counseling included regular oral hygiene, i.e. tooth brushing with fluoride-containing toothpaste twice a day, advice of a healthy diet with proper timing and composition of meals avoiding sugary snacks, and to use xylitol products on regular basis. Additionally, in the program of oral hygiene and fluoride, the parents were given counseling on how to brush their own teeth with fluoride-containing toothpaste and clean between them. In the program of diet and xylitol parent was asked to fill in one-day diary of his or her own diet in the waiting room, and the dental professional pointed out the frequency of meals and snacks, as well as suggested the use of xylitol 5 grams per day.

The children, accompanied by their parents, were clinically examined in various health clinics of the Vantaa public dental service. At the regular two-year visit, the dental hygienists and in-service trained dental nurses tested the children for mutans streptococci in plaque. The transtheoretical model and the motivational interviewing were introduced to the dental hygienists and in-service trained dental nurses to use in preventive counseling.

The results of this study will be published in three articles.

ELIGIBILITY:
Inclusion Criteria:

* first born children born in 2008

Exclusion Criteria:

* not first born children

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2008-01; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The colonization of mutans streptococci bacteria | At the age of 2 years
  The children were tested for the amount of mutans streptococci bacteria in their dental plaque at the age of 2 years. The recommended age for testing was 2-2.5 years, and the inclusion limits 2 years and 3 years.

SECONDARY OUTCOMES:
Dental caries | at the age of two
  At the age of two years, the children, accompanied by their parents, were clinically examined in the Vantaa PDS. The dental hygienists and in-service trained dental nurses that were working in each clinic performed the examinations by a mirror using the WHO criteria of the electronic patient database. The dental professionals were not blinded to the group of the child. The information from the clinical examinations, including the number of decayed teeth or teeth with distinct visual changes in enamel, was recorded on the database. No missed or filled teeth were found.

OTHER OUTCOMES:
Tooth brushing | At the age of two
  the habit of tooth brushing at the age of two years was asked by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kaisu Pienihäkkinen, docent, Study Director — University of Turku
Locations (1):
- Health and social and welfare affairs, oral health, Vantaa, Finland

IPD SHARING:
Plan to Share IPD: No
The individual participant data is not planned to be shared with other researchers, it will be destroyed after the study.

REFERENCES:
- [Result] Arpalahti I, Jarvinen M, Suni J, Pienihakkinen K. Acceptance of oral health promotion programmes by dental hygienists and dental nurses in public dental service. Int J Dent Hyg. 2012 Feb;10(1):46-53. doi: 10.1111/j.1601-5037.2011.00517.x. Epub 2011 Jun 23. PMID 21699653
- [Result] Arpalahti I, Tolvanen M, Pienihakkinen K. Comparing health promotion programs in public dental service of vantaa, Finland: a clinical trial in 6-36-month-old children. Int J Dent. 2013;2013:757938. doi: 10.1155/2013/757938. Epub 2013 Nov 18. PMID 24348559
- [Result] Arpalahti I, Jarvinen M, Kommonen HM, Tolvanen M, Pienihakkinen K. Parental Opinions on Children's Oral Health Counselling and Readiness to Change Health Habits. Oral Health Prev Dent. 2016;14(6):535-545. doi: 10.3290/j.ohpd.a37139. PMID 27957564
- [Derived] Arpalahti I, Hanninen K, Tolvanen M, Varrela J, Rice DP. The effect of early childhood non-nutritive sucking behavior including pacifiers on malocclusion: a randomized controlled trial. Eur J Orthod. 2024 Oct 1;46(5):cjae024. doi: 10.1093/ejo/cjae024. PMID 39119981
- See also: Doctoral thesis (article-based) — http://urn.fi/URN:ISBN:978-951-29-6180-1